CLINICAL TRIAL: NCT00634010
Title: Morphine Versus Methadone As First Line Strong Opioid for Cancer Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-0477; 1R01CA124481-01A1 (NIH); NCI-2012-02126 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Advanced Cancer; Solid Tumors
Keywords: Advanced Cancer; Solid Tumors; Cancer Pain; Opioid Pain Killer; Morphine; Methadone
MeSH Terms: conditions — Cancer Pain | interventions — Morphine; Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine Capsule (Active Comparator): Morphine 15 mg slow release orally every 12 hours + additional doses as needed
  Interventions: Drug: Morphine
- Methadone Capsule (Active Comparator): Methadone 5 mg orally every 12 hours + additional as needed doses up to 40-50 mg/day
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Morphine — 15 mg oral every 12 Hours; additional capsules taken every 2 hours as needed.
  Arms: Morphine Capsule
Drug: Methadone — 5 mg orally every 12 hours; additional capsules every 2 hours as needed.
  Arms: Methadone Capsule

SUMMARY:
Primary Aims:

* To determine whether methadone used as first line strong opioid is superior to morphine as evidenced by reduced pain over a 12-week treatment period in patients with advanced cancer. Previous studies have demonstrated consistent improvement of pain control after opioid rotation from morphine to methadone. In addition, the pilot study showed that there was a trend towards lower pain intensity when methadone used as first line opioid as compared to morphine. Researchers postulate that due to its superior analgesic effects, methadone will result in better pain control over time as compared to morphine.
* To determine whether methadone used as first line strong opioid is superior to morphine as evidenced by reduced frequency of neurotoxicity, dose escalation and treatment failure over a 12-week treatment period. Previous studies have demonstrated that patients develop increased pain or neurotoxicity after chronic use of morphine and require frequent opioid escalation. Researchers postulate that methadone will demonstrate lower opioid induced neurotoxicity, less frequent dose escalation and less treatment failure over 12-week treatment period as compared to morphine.

Secondary Aim:

-To perform an economic evaluation, comparing the costs and clinical benefits of methadone and morphine. Researchers will perform an evaluation that incorporates both treatment and potential "downstream" costs, as well as an examination of clinical benefits that incorporate preferences, to perform an appropriate economic comparison. We postulate that methadone and its associated costs will be cheaper than morphine. However, if one strategy is both more expensive and clinically superior than the other, researchers are prepared to perform an incremental cost-effectiveness analysis. In that case, researchers expect to show that the greater pharmaceutical costs involved with morphine will make its use not be a cost-effective strategy.

DETAILED DESCRIPTION:
STUDY DRUGS:

MORPHINE is recommended as the first choice of strong pain killers by the World Health Organization Pain Relief Guidelines.

METHADONE is recommended as the second choice of strong pain killers.

SCREENING TESTS:

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* You will be asked about your level of pain.
* You will be asked about any pain killers you are currently taking.
* You will be asked about your history of allergies.
* Blood (about 1 teaspoon) will be drawn to check your kidney function.

STUDY GROUPS:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of the coin) to 1 of 2 treatment groups. Group 1 will receive morphine while on-study. Group 2 will receive methadone. You will have an equal chance of being placed in either group. Neither you nor any of the study staff will know which study drug you are receiving. However, if needed for your safety, the study staff and study doctor will be able to find out which study drug you are receiving.

STUDY DRUG ADMINISTRATION:

If you are in Group 1, you will take 1 morphine capsule every 12 hours with water. If you are in Group 2, you will take 1 methadone capsule every 12 hours. Morphine and methadone should be swallowed whole.

You will be given additional capsules in another bottle to take for excessive pain. The additional capsules should be taken every 2 hours, as needed. If you need 3 or more of these additional doses in 24 hours, you should contact the study staff.

STUDY VISITS:

You will return to the clinic at the end of Weeks 1, 2, 4, 6, 8, 10 and 12 for questionnaires about your pain levels, ability to sleep, constipation, other side effects, and quality-of-life. You will complete 6 questionnaires at the Weeks 1, 2, 6, 10, and 11 visit. You will complete 11 questionnaires at the Weeks 4, 8, and 12 visits. Each questionnaire will take 1-3 minutes to complete. The visit with the research nurse will last about 45 minutes to 1 hour. Your study drug supply will also be checked. You also will be asked about your overall health, non-health care questions, and activity level. At these visits, you will receive a new prescription for a 2-week supply of the study drug.

PATIENT DIARY:

You will be given a patient diary booklet before you start taking the study drug. You will be asked to record when you take the study drug, other medications you may be taking, and any side effects you experience. You will fill out the patient diary once a day. It will take less than 2 minutes to complete.

For the first week of the treatment, you will be contacted by the research nurse every day either in person (if you are in the hospital) or by phone to check for pain, side effects, and the number of pills you have taken.

You are allowed to take other medication, such as medications for constipation, nausea, and other drugs during the study. All changes in medication for either symptoms or complications must be recorded by the research nurse at each study visit.

LENGTH OF STUDY:

After the visit at the end of Week 12, you will be off-study. You will be taken off-study early if your pain gets worse or intolerable side effects occur.

This is an investigational study. Both morphine and methadone are FDA approved and commercially available. You will not be told which study drug you were receiving. Up to 250 patients will take part in this study. Up to 200 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has pain caused by advanced cancer (local recurrence or metastatic disease)
2. Patient reporting average pain score for the last 24 hours is >/= 4 on a numerical scale from 0 to 10 (0= no pain, 10=the worst possible pain).
3. Patient is receiving mild opioids (e.g. propoxyphene, codeine, tramadol, hydrocodone), mixed agonist/antagonist (e.g. buprenorphine) or no opioids.
4. Patient requires initiation of strong opioid for cancer pain.
5. Patient has the ability to receive morphine or methadone orally.
6. Patient has no known allergy or severe toxicity to morphine or morphine-like drugs (e.g. hydromorphone, oxycodone, oxymorphone, codeine, hydrocodone, levorphanol), or methadone or methadone-like drug (e.g. propoxyphene).
7. Patient has normal cognition defined as normal state of arousal and absence of obvious clinical findings of confusion, memory or concentration deficit.
8. Patient has normal renal function (creatinine and blood urea nitrogen (BUN) within normal limits) </= 4 weeks of study entry.
9. Patient's performance status (ECOG) is 3 or less.
10. Patient is willing to sign written informed consent.
11. Patient is 18 years of age or older.
12. Patient is able to return to clinic for evaluation by physician day 8 , 15 , 29, 57 and 85 ( +/- 3 days) during study period.

Exclusion Criteria:

1. Patient has concurrent strong opioid for cancer pain, such as morphine, hydromorphone, oxycodone, meperidine, fentanyl, oral transmucosal fentanyl citrate (OTFC), sufentanil, methadone, levorphanol, transdermal fentanyl.
2. Patient is receiving radiation therapy for pain control.
3. Patient is receiving drugs that interacting with methadone, such as (delavirdine, fluconazole, fluvoxamine, bravavir, amprenavir, efavirenz, lopinavir, nelfinavir, nevirapine, carbamazepine, dexamethasone (Patients receiving short term chemotherapy-related doses are permitted) , phenytoin, rifampin, or grapefruit,).
4. Patients are determined incapable of completing the evaluation forms.
5. Severe hypotension, acute or severe asthma, paralytic ileus, gastrointestinal obstruction, severe respiratory depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - LBJ General Hospital, Houston, Texas
  - The Michael E. DeBakey V.A. Medical Center, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: February 22, 2008 to September 14, 2010. All recruitment done within medical clinics at The University of Texas MD Anderson Cancer Center and Lyndon Baines Johnson Hospital.
Groups:
- Morphine Capsule: Morphine 5 mg slow release morphine orally every 12 hours and 5 mg immediate-release morphine every 2 hours as needed for breakthrough pain.
- Methadone Capsule: Methadone 5 mg orally every 12 hours and 5 mg immediate-release (IR) Morphine every 2 hours as needed for rescue pain (for first week).
Period: Overall Study
Arm/Group | Morphine Capsule | Methadone Capsule
Started | 18 | 18
Completed | 8 | 4
Not Completed | 10 | 14
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Disease Progression | 1 | 1
Not completed — Non-Compliant | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine Capsule | Methadone Capsule | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.00 (8.677) | 60.39 (12.069) | 57.4 (10.430)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Participant Pain Severity Score Measured Using Brief Pain Inventory
Description: Brief Pain Inventory (BPI): Pain severity measured with BPI, which asks participants to rate pain for last 24 hours on 0 to 10 scales at its "worst", "least", "average " and "now". The scales are presented on a 10 cm line, with each number equidistant from the next. Each scale is bounded by the words "no pain' at the 0 end and "pain as bad as you can imagine" at the other. BPI used to determine whether methadone used as first line strong opioid is superior to morphine as evidenced by reduced pain over a 4 week (+/- 3 days) treatment period in participants with advanced cancer.
Time Frame: Comparing baseline and pain scores at 4 weeks (+/- 3 days)
Population: The study was terminated without completing any analysis because the sample size was too small to detect any differences between the groups. Participants eligible for the study often had significant symptom distress and could not continue in the four week study period needed for data collection contribution to mean calculation.
Arm/Group | Morphine Capsule | Methadone Capsule
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from baseline to Day 85, anticipated study period 12 weeks.
Arm/Group | Morphine Capsule | Methadone Capsule
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 13/18 | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Capsule (N=18) | Methadone Capsule (N=18)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (10) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (3)
Alkaline phosphatase increased (Investigations) | 2 (2) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 4 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (4) | 0 (0)
Atrophy skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (29)
Bilirubin increased (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (5) | 2 (3)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Cardiac troponin T increased (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (10) | 5 (7)
Constipation (Gastrointestinal disorders) | 11 (37) | 12 (30)
Creatinine increased (Investigations) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 5 (5) | 9 (20)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 6 (15)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 6 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (8)
Edema limbs (General disorders) | 4 (4) | 6 (10)
Esophageal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (2) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (4)
Fatigue (General disorders) | 8 (8) | 11 (32)
Fever (General disorders) | 1 (1) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Hemoglobin decreased (Metabolism and nutrition disorders) | 4 (16) | 2 (4)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection (Other) (Infections and infestations) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 6 (9) | 4 (11)
Leukopenia (Investigations) | 2 (11) | 2 (3)
Metabolic/Laboratory (Other) (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (37) | 11 (29)
Neurology (Other) (Nervous system disorders) | 2 (10) | 2 (5)
Neutrophil count decreased (Investigations) | 1 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (3) | 2 (2)
Pain (General disorders) | 2 (4) | 0 (0)
Pain (Other) (General disorders) | 3 (5) | 10 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (57) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Psychiatric disorders) | 2 (3) | 4 (8)
Personality change (Psychiatric disorders) | 1 (2) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (6) | 3 (5)
Serum cacium decreased (Metabolism and nutrition disorders) | 2 (4) | 2 (2)
Serum glucose decrease (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (4) | 2 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (4) | 1 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (6) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 3 (8)
Taste alteration (Nervous system disorders) | 0 (0) | 3 (3)
Thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Ureteric hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (10) | 5 (12)
Watering eyes (Eye disorders) | 0 (0) | 1 (2)
Weight loss (Investigations) | 1 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes